CLINICAL TRIAL: NCT03837379
Title: Development and Testing of a Depression-Specific Behavioral Activation Mobile App Paired With Nicotine Replacement Therapy Sampling for Smoking Cessation Treatment Via Primary Care
Brief Title: Goal2Quit + NRT Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Dahne, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00074015; K23DA045766 (NIH)
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Cigarette Smoking; Smoking Cessation; Depression
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation; Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (Other): Participants in the Treatment As Usual condition will receive educational material on quitting smoking. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Interventions: Behavioral: Treatment as Usual
- Goal2Quit + NRT Sampling (Experimental): Participants in the Goal2Quit + NRT Sampling condition will receive a download code to download the Goal2Quit mobile application. Goal2Quit is a mobile app for cigarette smokers with elevated symptoms of depression. Within the app, users identify values, create activities, schedule activities, rate mood daily, and track cigarette smoking. Participants in Group B will also receive a two-week "starter kit" sample of nicotine replacement therapy (NRT; 14mg patch and 4mg lozenge). Participants will be asked to utilize Goal2Quit regularly, at least once per day, as well as the NRT sample in an attempt to quit smoking. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Interventions: Combination Product: Goal2Quit + NRT Sampling

INTERVENTIONS:
Behavioral: Treatment as Usual — Participants in the Treatment As Usual condition will receive educational material on quitting smoking. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Arms: Treatment As Usual
Combination Product: Goal2Quit + NRT Sampling — Participants in the Goal2Quit + NRT Sampling condition will receive a download code to download the Goal2Quit mobile application. Goal2Quit is a mobile app for cigarette smokers with elevated symptoms of depression. Within the app, users identify values, create activities, schedule activities, rate mood daily, and track cigarette smoking. Participants in Group B will also receive a two-week "starter kit" sample of nicotine replacement therapy (NRT; 14mg patch and 4mg lozenge). Participants will be asked to utilize Goal2Quit regularly, at least once per day, as well as the NRT sample in an attempt to quit smoking. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Arms: Goal2Quit + NRT Sampling

SUMMARY:
The goal of this work is to develop, systematically evaluate, and clinically test an integrated cessation intervention comprised of a depression-specific Behavioral Activation (BA) for cessation mobile app ("Goal2Quit") packaged with nicotine replacement therapy (NRT) sampling. This integrated intervention will address the need for an easily disseminable, evidence-based, depression-specific cessation intervention for delivery via primary care.

ELIGIBILITY:
Inclusion Criteria:

* Current elevated depressive symptoms defined as a score of > 10 (at least mild depression) on the Patient Health Questionnaire-8 (PHQ-8)
* Current smoking, defined as smoking 10+ cigarettes/day, for 25+ days out of the last 30, for the last 6+ months
* Ownership of an Android or iOS smartphone
* Age 18+
* Possess a valid e-mail address that is checked daily to access follow-up assessments
* English fluency

Exclusion Criteria:

- Contraindications for NRT (pregnancy/intention to become pregnant/breastfeeding, recent cardiovascular trauma/uncontrolled hypertension) - Severe visual impairment, which may limit ability to utilize an app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dahne, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahne J, Wahlquist AE, Kustanowitz J, Natale N, Fahey M, Graboyes EM, Diaz VA, Carpenter MJ. Behavioral Activation-Based Digital Smoking Cessation Intervention for Individuals With Depressive Symptoms: Randomized Clinical Trial. J Med Internet Res. 2023 Nov 1;25:e49809. doi: 10.2196/49809. PMID 37910157

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment As Usual | Goal2Quit + NRT Sampling
Started | 50 | 114
Completed | 47 | 103
Not Completed | 3 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment As Usual | Goal2Quit + NRT Sampling | Total
Number analyzed (Participants) | 47 | 103 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (11.2) | 37.1 (9.7) | 38.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 53 | 80
  Male | 20 | 50 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 13
  Not Hispanic or Latino | 43 | 94 | 137
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 21 | 33
  White | 26 | 74 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: 7 Day Point Prevalence Abstinence
Description: Patients will self report smoking status (yes/no) for the seven days preceding the 12-week follow-up assessment. The data reported is based on the participants that reported yes.
Time Frame: From 7 days preceding the 12-week follow-up assessment through the 12-week follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | Goal2Quit + NRT Sampling
Number analyzed (Participants) | 47 | 103
Participants | 1 | 16

2. Secondary Outcome: Mean Score of Depressive Symptoms
Description: Patients will self report depressive symptoms weekly for 8 weeks with final follow-up at 12-weeks via the Beck Depression Inventory-II. The range of scores possible are 0 - 63, where lower scores are indicative of lower symptoms of depression.
Time Frame: Change in BDI from baseline to Week 12
Population: The overall number of participants analyzed is inconsistent because this is the number of participants that completed their week 12 surveys in order to be included in this particular data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment As Usual | Goal2Quit + NRT Sampling
Number analyzed (Participants) | 34 | 66
score on a scale | -6.97 (11.15) | -9.06 (11.60)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment As Usual | Goal2Quit + NRT Sampling
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/103
Other Adverse Events (participants affected / at risk) | 0/47 | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT03837379/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT03837379/ICF_000.pdf